CLINICAL TRIAL: NCT02002091
Title: Prevalence of Micro and Macroangiopathy in Newly Diagnosed type2 Diabetic Adults in Suburban Area of Algiers
Brief Title: Morbidity in Newly Diagnosed type2 Diabetes in Adults
Acronym: MORNDIAB
Status: Completed | Type: Observational
Sponsor: University of Algiers (Other)
Collaborators: National Institute of public Health, Algeria (Unknown); Hopital Ain Taya (Other); Parnet Hospital (Other); Hôpital Mustapha Pacha (Other); Birtraria Hospital (Other); Bab El Oued Teaching Hospital (Other)
Responsible Party: Principal Investigator, W.N. Nibouche-Hattab, Assistant Professor, University of Algiers
Other Study IDs: UAlgiers FM 401/desm/07
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Type2 Diabetes Mellitus; Complications
Keywords: Type2 diabetes mellitus; Microangiopathy; Chronic Kidney disease; Cardiovascular disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood. Urines. Tissue (kidney) for few patients.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Complications,no specific treatment: After screening for complications, a non specific multi interventional treatment is applied to patients. After one year of follow up, we will compare two groups: with and without chronic kidney disease, on the advent of cardiovascular events. An adjustment is done for age and major risk factors.
  Interventions: Other: no specific treatment

INTERVENTIONS:
Other: no specific treatment — lifestyle counseling, antihypertensive drugs, antidiabetic drugs (oral and / or insulin)treatment of comorbidity or complications of diabetes.

SUMMARY:
* It is a prospective,observational, cohort study
* The main purpose of the study is to assess the prevalence of diabetic chronic complications in newly diagnosed type 2 diabetics in suburban area of Algiers.
* The secondary purpose is to study the impact of diabetic renal complications as a risk factor on the atherothrombotic events.

DETAILED DESCRIPTION:
To reach the two purposes, we need to conduct a cohort study:

* The cohort population is type 2 diabetes patients that have been recruited in a consecutive and exhaustive way. The first consultation is performed in hospital or in one of 12 primary care units of Ain-Taya's health sector in Est suburb of Algiers . When a glycemia is found at 1.26 g/litre or over, the patient is referred to principal investigator to confirm the diagnosis of type 2 diabetes ,to recruit him and proceed to complete screening for chronic complications
* For the main purpose, we evaluate the prevalence of micro and macrovascular complications, at the time of diagnosis, in type2 diabetes patients that have been recruited. For some complications as Diabetic Kidney Disease, we have to follow up the patient at least three months to confirm the chronic nature of the nephropathy.
* For the secondary purpose, the cohort population is followed up for one year, the patients are treated commonly. We'll check out all the cardiovascular events linked to atherothrombosis.Two groups of patients might be formed:

  * The first group is composed of all diabetic patients, with chronic Kidney disease (CKD) and without atherothrombotic disease. CKD is defined by albuminuria (micro or macroalbuminuria) and/or renal failure, present for more than 3 months . All the patients with CKD are considered to be "exposed" to atherothrombotic disease.
  * The second group is composed of all diabetic patients, without CKD and without atherothrombotic disease. This group is considered to be "not exposed" to the atherothrombotic disease.

We will compare the two groups, on occurence of cardiovascular events, after adjustment of age and major cardiovascular risk factors, and after excluding patients 'not exposed' having had a prior treatment with conversion enzyme inhibitor or angiotensin receptor antagonist .

* The size of the sample is calculated with statistical formula:

  n= E2 Po Qo / i2 n= size of the sample E= 1.96 with error risk : alpha= 5% Po= 30% Qo= 1-Po "n" is at least egal to 323 patients
* Statistical analysis is performed with epi info 6.04b and all tests are performed with an error risk alpha= 5%

  * Descriptive statistics of patients characteristics:

    * For quantitative variables,we will calculate means,standard deviations, median and quantiles.
    * for qualitative variables, percentage will be calculated.
  * Comparative statistics according to existence of renal disease or not

    * Khi-square test is performed for qualitative variables
    * Student test: for two means comparison
    * Anova test: to compare more than two means
  * Multivariate analysis will be done on SPSS v: 21 software program, adjustment will be done for age, sexe and major cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged from 40 to 70 years
* Newly diagnosed type 2 diabetes
* Never treated for diabetes

Exclusion Criteria:

* Gestational diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of type 2 diabetes patients that diabetes is diagnosed recently, in one of the health structures, in the east suburban area of Algiers. In the first step they are recruited by primary care physicians, on the basis of glycemia >= 1.26 g/l (capillary or venous); then they are automatically directed to the main investigator, in hospital consultation, to confirm by two blood samples, the hyperglycemia; and (second step) screen for differential diagnosis (secondary diabetes)before the definitive recruitment.Patients are systematically,consecutively recruited. They are followed up during 1 year, they are seen every 3months at least.
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Biad, professor, Study Director — University of Algiers -Faculté de Medecine-; Wafia-Nadia Nibouche- Hattab, Ass-Prof, Principal Investigator — University of Algiers -Faculté de Médecine-
Locations (1):
- Internal Medicine department - Ain-Taya's Hospital, Aïn Taya, Algiers Province, Algeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nibouche WN, Biad A. [Arterial hypertension at the time of diagnosis of type 2 diabetes in adults]. Ann Cardiol Angeiol (Paris). 2016 Jun;65(3):152-8. doi: 10.1016/j.ancard.2016.04.017. Epub 2016 May 24. French. PMID 27234335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 327 patients aged from 40 to 70 years were seen from 2009 to 2013. The main investigator confirmed the diagnosis of type 2 diabetes. A secondary diabetes was excluded before definitive recruitment. When the diagnosis of type 2 diabetes is highly probable and ensure that it was newly diagnosed, we screened for all chronic complications.
Groups:
- Complications' Assessment for Men: 122 patients had a complete clinical examination, we realized an electrocardiogram, some biological exams for glycemic, hepatical, hematological and inflammatory status. We performed, in assessing macroangiopathy, an echocardiography, a vascular ultrasonography, a cardiac stress testing ( myocardial scintigraphy or stress electrocardiogram), a coronaroangiography if indicated and a cerebral scanner in case of suspicion of stroke. For the assessment of microangiopathy, we practiced a fundoscopy, a neurological examination to screen for peripheral neuropathy in all patients, we performed the Ewing tests for cardiac autonomic neuropathy , post voiding residual for diabetic cystopathy, a manocystometry if indicated and evaluated the renal status (ACR, creatininemia, uro-nephrological echography) in all patients.
- Complications' Assessment for Women: 205 patients had a complete clinical examination, we realized an electrocardiogram, some biological exams for glycemic, hepatical, hematological and inflammatory status. We performed, in assessing macroangiopathy, an echocardiography, a vascular ultrasonography, a cardiac stress testing (myocardial scintigraphy or stress electrocardiogram) to screen for ischemic myocardial, a coronaroangiography if indicated and a cerebral scanner in patients with suspected stroke. For the assessment of microangiopathy, we practiced a fundoscopy by an ophtalmologist, a neurological examination to screen for peripheral neuropathy, we performed the Ewing tests to screen for cardiac autonomic neuropathy, a post voiding residual to search for diabetic cystopathy, a manocystometry if indicated and evaluate the renal status (ACR, creatininemia, uro-nephrological echography) in all patients.
Period: Screening
Arm/Group | Complications' Assessment for Men | Complications' Assessment for Women
Started | 122 | 205
Completed | 109 | 191
Not Completed | 13 | 14
Not completed — Lost to Follow-up | 10 | 12
Not completed — Death | 3 | 2
Period: One Year Follow up
Arm/Group | Complications' Assessment for Men | Complications' Assessment for Women
Started | 109 | 191
Completed | 109 | 191
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We described gender, age, history of familial, major cardiovascular risk factors and mean anthropometric, blood pressure and biological measures
Groups:
- Men Population: Screening for all chronic complications were performed for men. A non specific multi interventional treatment is applied to patients, as lifestyle counseling, antihypertensive drugs, antidiabetic drugs (oral and / or insulin) treatment of comorbidity or complications of diabetes as soon as the patients are recruited.
- Women Population: Screening for all chronic complications were performed for women. A non specific multi interventional treatment is applied to patients, as lifestyle counseling, antihypertensive drugs, antidiabetic drugs (oral and / or insulin)treatment of comorbidity or complications of diabetes as soon as the patients are recruited.
- Total: Total of all reporting groups
Arm/Group | Men Population | Women Population | Total
Number analyzed (Participants) | 122 | 205 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.9) | 53.7 (8.4) | 53.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 205 | 205
  Male | 122 | 0 | 122
Region of Enrollment [Number; unit: participants]
  Algeria | 122 | 205 | 327
history of family diabetes [Number; unit: participants] | 84 | 138 | 222
history of family hypertension [Number; unit: participants] | 69 | 133 | 202
waist circumference [Mean (Standard Deviation); unit: cm] | 98.1 (10.4) | 99.3 (10.8) | 98.9 (10.7)
BMI [Mean (Standard Deviation); unit: kg/m²] | 26.6 (4.9) | 28.9 (5.1) | 28.0 (5.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 139.9 (22.6) | 141.9 (23.9) | 141.2 (23.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 86.6 (13.0) | 85.3 (10.9) | 85.8 (11.7)
Glycaemia [Mean (Standard Deviation); unit: g/l] | 2.70 (1.05) | 2.39 (0.98) | 2.50 (1.01)
glycated hemoglobin [Mean (Standard Deviation); unit: percent] | 9.73 (2.16) | 9.48 (2.38) | 9.58 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Number and Prevalence of Patients With Diabetic Retinopathy
Description: * Conventional ophtalmoscopy has been used to screen for diabetic retinopathy by an ophtalmologist at his office.
  * Retinal angiography was performed if indicated by the ophtalmologist
Time Frame: At recruitment
Population: From 327, 309 (113 men and 196 women) patients benefit from ophthalmoscopy with a trained ophthalmologist. 18 patients (9 men and 9 women) didn't perform the test. Each patient having a diabetic retinopathy was treated by the ophtalmologist who performed the examination
Measure: Count of Participants; unit: Participants
Groups:
- Men Group; Women Group: Patients were assessed for diabetic retinopathy.
Arm/Group | Men Group | Women Group
Number analyzed (Participants) | 113 | 196
Participants | 9 | 18
Statistical Analysis 1: Comparison: Men Group vs Women Group; Test type: Other; p = 0.706, Chi-squared

2. Primary Outcome: Number of Patients With Distal Diabetic Neuropathy
Description: All 327 patients had a neurological examination by the same physician to screen for Distal Diabetic Neuropathy:
  * Distal sensory testing: including 10 g monofilament test, vibration perception with 128 Hz tuning fork, temperature, touch , prickling and pain perception
  * Ankles and knees reflex testing
  * Muscle strength testing (quadriceps and tibialis anterior)
  * We use the Michigan Neuropathy Screening Instrument score. We consider the diagnosis of Distal Diabetic Neuropathy if the score is up of 2 in at least one food. The MNSI score is ranged from 0 to 5 for each food
  * Use of neuropathic pain score (DN4), if the DN4 is found up or egal to 4 we consider the diagnosis of neuropathic pain. The DN4 score is ranged from 0 to 10
Time Frame: At recruitment
Population: We exclude from analysis 10 patients (2 men and 8 women) with neuropathy because of other possible etiology (8 hypothyroidism, 1 with B12 deficiency,1 with narrowed lumbar vertebra channel)
Measure: Count of Participants; unit: Participants
Groups:
- Men Group: All 122 patients were examined twice with the same method by the same physician.
- Women Group: All 205 women were examined twice by the same physician that had examined men with the same method
Arm/Group | Men Group | Women Group
Number analyzed (Participants) | 120 | 197
Participants | 42 | 56
Statistical Analysis 1: Comparison: Men Group vs Women Group; Test type: Other; p = 0.346, Chi-squared

3. Primary Outcome: Number of Patients With Chronic Kidney Disease (CKD)
Description: * We screened for albuminuria or microalbuminuria in 24h urine collection with turbidimetry or immuno turbidimetry method ( performed 3 times in 4 or 6 months )
  * Measurement of albumine- to- creatinine ratio (ACR), Albuminuria was diagnosed if ACR > or egal to 30 mg/g at least twice in 4 to 6 months. We ensure before performing ACR that there was no dysglycaemia, no urinary infection, no fever nor forced diuresis before we evaluate the urine sample.
  * Cyto bacteriological examination and urine culture
  * Serum creatinine repeated 2 to 3 time within 4 to 6 months
  * Glomerular filtration rate was assessed with the Modification of Diet in Renal disease study equation (MDRD)
  * Renal and urine tract echography to measure the kidneys and to screen for urine tract dilatation We made the diagnosis of Chronic Kidney Disease (CKD) if the glomerular filtration rate was < 60 ml/min/1.73 m² and/or ACR > or equal to 30 mg/g with a permanent character
Time Frame: At recruitment
Population: Of 327 patients, 317 had a complete screening for chronic kidney disease, 5 men and 5 women were excluded from analysis because of incomplete renal status.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: Screening for chronic kidney disease have been made for all patients.
- Women Group Population: Screening for chronic kidney disease was performed in all patients.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 117 | 200
Participants | 35 | 43
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Other; p = 0.123, Mantel Haenszel

4. Primary Outcome: Number of Patients With Hypertension
Description: * Blood pressure measurement by electronic tensiometer (OMRON 3 or 4) on the right and left arm, after 10 mn of supine position.
  * Three measures were performed with respect of one minute interval between each measure.
  * Mean blood pressure is calculated
  * Three other measures are performed in Three ulterior consultations
  * Hypertension is diagnosed if the mean blood pressure >= 140 /90 mm Hg
Time Frame: At recruitment
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: Hypertension was screened in patients at the time of diagnosis of type 2 diabetes. 19 patients already had hypertensive drugs.
- Women Group Population: Hypertension was screened in all women in the same conditions than men. 49 patients had antihypertensive drugs.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 122 | 205
Participants | 82 | 136
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Other; p = 0.968, Chi-squared, Corrected

5. Primary Outcome: Number of Patients With Silent Myocardial Ischemia
Description: * 9 derivations resting electrocardiogram (ECG)
  * Echocardiography
  * Standard ECG stress test
  * Stress Myocardial Perfusion scintigraphy if patients are not able to perform ECG stress test
  * Coronary angiography if the exercise ECG stress test or stress myocardial perfusion scintigraphy suggest high probability of coronary heart disease
Time Frame: At recruitment
Population: 88.9 % (291 patients) had a screening for coronary heart disease. We performed an electrocardiogram in 325 cases, an echocardiography in 317 cases, a myocardial ischemic test in 291 cases (223 for silent myocardial ischemia: 85 men and 138 women) and a coronarography in 18 cases ( 8 men and 10 women, all had a positive myocardial ischemic test)
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: We screened for silent myocardial ischemia . We ensure of the absence of a chest pain in patients we screened.
- Women Group Population: We screened for silent myocardial ischemia in 138 asymptomatic patients.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 85 | 138
Participants | 11 | 4
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.004, Fisher Exact — The threshold for statistical significance for P-Value is <0.05

6. Primary Outcome: Number of Patients With Lower Extremity Artery Disease
Description: * Search for history of intermittent claudication
  * Complete vascular examination with Ankle-Brachial Index (ABI) measurement.
  * Lower limb duplex ultrasonography.
Time Frame: At recruitment
Population: Lower limb duplex ultrasonography measurement has been done in 306 among 327 patients (111 men and 195 women). 21 patients, with a lack of data,were excluded from analysis. Chi 2 test was used for comparison of proportions.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: In the men's group screened for lower limb arterial disease, there were significantly more tobacco use (52 patients) than in the women's group (see characteristics)
- Women Group Population: In the women's group 33 patients had a tobacco use
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 111 | 195
Participants | 6 | 12
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.988, Fisher Exact

7. Primary Outcome: Number of Patients With Carotid Artery Stenosis
Description: * Screening for carotid murmur at clinical examination by the same physician for all patients
  * Carotid duplex ultrasonography with intima-media thickness measurement. All atherosclerotic lesions were reported.
Time Frame: At recruitment
Population: From 327, 304 patients (109 men and 195 women) could perfom duplex ultrasonography of supra aortic trunks. We focus on the examination of external and internal carotids.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: The men's group had some characterictics that differ from women's group. Tobacco is more widely used in men
- Women Group Population: The women in this group have a mean body mass index higher than in the men's group
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 109 | 195
Participants | 7 | 3
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.038, Fisher Exact

8. Primary Outcome: Number of Patients With Renal Artery Stenosis or Elevated Intrarenal Resistance Index
Description: - Renal artery duplex ultrasonography has been performed only if the patient presents a resistant hypertension treated with four drugs, including a diuretic or if blood pressure was over 180/10 mm Hg at recruitement.
Time Frame: At recruitment
Population: From 327 we perform a duplex ultrasonography of renal arteries in 16 patients (6 men and 10 women) The number of participants analyzed is too small to have a statistical analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: Those patients who perform renal artery ultrasonography had severe hypertension treated with at least four anti hypertensive drugs including one diuretic or a blood pressure over 180/100 mm Hg
- Women Group Population: Patients that had an ultrasonography of renal arteries, had severe hypertension treated with at least four anti hypertensive drug including one diuretic or a blood pressure over 180/100 mm Hg
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 9 | 10
Participants | 2 | 2

9. Primary Outcome: Number of Patients With Cardiac Autonomic Neuropathy
Description: * Conditions of the Ewing tests: fasting, resting at least 30mn, no hypoglycemia and no effort within 24hours, no drugs that interfere with heart rate.
  * Ewing Tests for cardiac autonomic neuropathy: Beat-to-Beat heart rate variation, Heart rate response to standing, Heart rate response to valsalva maneuver, Systolic blood pressure response to standing. All tests have been performed with the same physician and aid
Time Frame: at recruitment
Population: We screened 283 patients from 327 (100 men and 183 women). We excluded 44 patients from analysis (22 men and 22 women)cause of beta blocker treatment or high blood pressure, or diabetic retinopathy, or severe coronary heart disease and patients that could not perform deep breathing.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: We screened the men's group for cardiac autonomic neuropathy.
- Women Group Population: .We screened women's group for cardiac autonomic neuropathy.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 100 | 183
Participants | 10 | 19
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.917, Chi-squared, Corrected

10. Primary Outcome: Number of Patients With Bladder Autonomic Neuropathy
Description: * History of recurrent urine tract infection and/or dysuria and/or incomplete bladder emptying
  * Post voiding residual(PVR) measurement with abdominal echography by a radiologist
  * Cystomanometry is performed if PVR > 50 ml
  * In men the prostatic measurement was made in all patients. In women, we measured the volume of uterus.
Time Frame: at recruitment
Population: From 327 we could screen 318 patients (118 men and 200 women) for bladder autonomic neuropathy. We performed a cystomanometry in 4 patients. We exclude, from analysis, 9 patients who didn't come to perform the post-voiding volume measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: In the men's group, the diagnosis of autonomic neuropathy of bladder was made as specified.
- Women Group Population: women were slightly older than men. the diagnosis was done the same way than in men.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 118 | 200
Participants | 5 | 11
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.816, Chi-squared, Corrected

11. Primary Outcome: Number of Patients With Gastro-intestinal Autonomic Neuropathy
Description: * We interviewed all patient, looking for a history of post prandial discomfort or bad gastric emptying sensation or vomiting or unexplained diarrhea or constipation
  * We performed an endoscopic examination to exclude other causes in patients with a positive history of gastro-intestinal troubles.
Time Frame: at recruitment
Population: An endoscopic examination has been performed in six women whose report vomiting, nausea or constipation. In the men's group no-one had an endoscopic examination.
Measure: Count of Participants; unit: Participants
Groups:
- Men's Group Population: All men participated to interview.
- Women Group Population: All women participated to interview.
Arm/Group | Men's Group Population | Women Group Population
Number analyzed (Participants) | 122 | 205
Participants | 0 | 6
Statistical Analysis 1: Comparison: Men's Group Population vs Women Group Population; Test type: Superiority or Other; p = 0.008, Fisher Exact — Statistical significance : p< 0.05

12. Primary Outcome: Number of Patients With Erectile Dysfunction
Description: - Questionary: onset , drug use, medical history, psycho- social conditions
Time Frame: at recruitment
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: 122 men were assessed for erectile dysfunction .
Arm/Group | Men Group Population
Number analyzed (Participants) | 122
Participants | 63

13. Secondary Outcome: Number of Patients With New Cardiac Events During Follow-up
Description: * We Record every documented acute coronary syndrome during follow-up;
  * Each patient had an electrocardiogram every 3 months and during acute cardiovascular events;
  * Echocardiography has been performed if indicated by the cardiologist.
Time Frame: One year after recruitment
Population: 305 patients (112 men and 193 women) were re-evaluated one year after recruitment. From 327 patients enrolled, we excluded 22 patients (10 men and 12 women) from the analysis because of a lack of data, they were lost from follow-up. We include in analysis 5 patients who died the three first months during follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: We re-evaluated all patients for cardiac events during one year after recruitment.
- Women Group Population: All women were re-evaluated during one year of follow-up.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 112 | 193
Participants | 7 | 2
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Other; p = 0.025, Chi-squared, Corrected — The threshold of statistical difference is P-value < 0.05

14. Secondary Outcome: Number of Patients With New Stroke or Transient Ischemic Attack
Description: * We assessed every new clinical signs of stroke with an interview searching for acute neurological symptoms and a clinical examination for all patients, from day one of recruitment to one year of follow-up;
  * Tomodensitometry if there was a clinical presentation of stroke. Magnetic resonance imaging if transient ischemic attack was suspected.
Time Frame: One year after recruitment
Population: 300 patients (109 men and 191 women) were re-evaluated one year after recruitment. From 327 patients enrolled, we excluded 27 patients (13 men and 14 women) from the analysis because of a lack of data. 22 patients (10 men and 12 women) were lost from follow-up and 5 died too early during follow-up (three first months).
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: All men were evaluated for stroke one year after recruitment.
- Women Group Population: All women were evaluated for stroke after one year of follow-up.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 109 | 191
Participants | 1 | 2

15. Secondary Outcome: Number of Patients With Lower Limbs Atherothrombotic Accident
Description: During one year of follow-up :
  * We search for a recent history of intermittent claudication;
  * We perform a systematic clinical examination with palpation of lower limb pulses and an Ankle-Brachial Index measurement after one year or in the presence of an acute ischemic lower limb episod ;
  * Lower limb duplex sonography in the presence of an abnormal clinical vascular examination;
  * Angiography in the presence of a lower limbs vascular event.
Time Frame: One year after recruitment
Population: 300 patients (109 men and 191 women) were re-evaluated one year after recruitment. From 327 patients enrolled, we excluded 27 patients (13 men and 14 women) from the analysis because of a lack of data, 22 patients (10 men and 12 women) were lost from follow-up and 5 died too early during follow-up (three first months).
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: 109 men were evaluated for new lower limb atherothrombotic events, after one year after recruitment.
- Women Group Population: 191 women were evaluated for lower limb atherothrombotic events, after one year of follow-up.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 109 | 191
Participants | 0 | 1

16. Secondary Outcome: Number of Patients That Died From Cardio Vascular Cause
Description: - We recorded each death and its cause from a medical record after hospitalization in emergency units or phone contact with the patient's relatives to have some news. The record began with recruitment.
Time Frame: One year after recruitment
Population: From 327 patients (122 men and 205 women) enrolled, 305 were followed-up one year or until death (112 men and 193 women). 22 patients (10 men and 12 women) were excluded from analysis because lost during follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Men Group Population: 112 men were evaluated and followed-up after recruitment.
- Women Group Population: 193 women were evaluated and followed-up from recruitment.
Arm/Group | Men Group Population | Women Group Population
Number analyzed (Participants) | 112 | 193
Participants | 3 | 2
Statistical Analysis 1: Comparison: Men Group Population vs Women Group Population; Test type: Other; p = 0.059, Fisher Exact — the threshold for statistical significance used is P-value <0.05

ADVERSE EVENTS:
Time Frame: One year after, adverse events were collected. We mean by adverse events all events, that disrupted during one year of follow-up, related to a non-specific treatment or to any pathological state or related or not to diabetic complications.
Description: During follow-up, we put in place a monitoring of any new clinical sign or biological change (renal or hepatic function). An assessment is performed regarding the new clinical or biological change.
Groups:
- Men's Group: From 122 men at recruitment, 112 had been followed-up one year or until death. 109 had complete one year of follow-up.
- Women's Group: From 205 women, 193 had been followed-up one year or until death. 191 women had complete one year of follow-up.
Arm/Group | Men's Group | Women's Group
All-Cause Mortality (participants affected / at risk) | 4/112 | 4/193
Serious Adverse Events (participants affected / at risk) | 3/109 | 4/191
Other Adverse Events (participants affected / at risk) | 18/109 | 29/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Men's Group (N=109) | Women's Group (N=191)
Atherothrombotic event (Vascular disorders) | 3 (4) | 4 (4) — Acute coronary syndrome Lower-limb acute arterial thrombosis Acute cerebrovascular event
OTHER ADVERSE EVENTS (reported when occurring in more than 0.016% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Men's Group (N=109) | Women's Group (N=191)
Moderate acute renal insufficiency (Renal and urinary disorders) | 3 | 4 — Rise of creatinine from the baseline, > 1.5 x or Glomerular filtration rate < 60 ml/min/1,73m²
New onset of permanent hypertension (Vascular disorders) | 15 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes